CLINICAL TRIAL: NCT04550832
Title: A Phase IIb, Open Label, Randomized Controlled Dose Ranging Multi-Center Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Exposure-Response Relationship of Different Doses of Delpazolid in Combination With Bedaquiline Delamanid Moxifloxacin in Adult Subjects With Newly Diagnosed, Uncomplicated, Smear-Positive, Drug-sensitive Pulmonary Tuberculosis
Brief Title: PanACEA DElpazolid Dose-finding and COmbination DEvelopment (DECODE)
Acronym: DECODE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Radboud University Medical Center (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCB01-0371-20-2-02; PanACEA-DECODE-01 (Other: PanACEA)
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Infections and Infestations; Pulmonary Tuberculosis
Keywords: drug-sensitive TB
MeSH Terms: conditions — Infections; Tuberculosis, Pulmonary | interventions — delpazolid; bedaquiline; OPC-67683; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm1(D0) (Active Comparator): Participants receive the following medication for the duration of 16weeks together with food.
  * Delpazolid : Will not administered
  * Bedaquiline: will be dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid: will be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin: will be dosed as per the licensed dose: 400 mg orally once daily
  Interventions: Drug: Bedaquiline, Delamanid, Moxifloxacin
- Arm2(D400) (Experimental): Participants receive the following medication for the duration of 16weeks together with food.
  * Delpazolid : Will be dosed 400 mg orally once daily
  * Bedaquiline: will be dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid: will be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin: will be dosed as per the licensed dose: 400 mg orally once daily
  Interventions: Drug: Delpazolid; Drug: Bedaquiline, Delamanid, Moxifloxacin
- Arm3(D800-OD) (Experimental): Participants receive the following medication for the duration of 16weeks together with food.
  * Delpazolid : Will be dosed 800 mg orally once daily
  * Bedaquiline: will be dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid: will be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin: will be dosed as per the licensed dose: 400 mg orally once daily
  Interventions: Drug: Delpazolid; Drug: Bedaquiline, Delamanid, Moxifloxacin
- Arm4(D1200) (Experimental): Participants receive the following medication for the duration of 16weeks together with food.
  * Delpazolid : Will be dosed 1200 mg orally once daily
  * Bedaquiline: will be dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid: will be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin: will be dosed as per the licensed dose: 400 mg orally once daily
  Interventions: Drug: Delpazolid; Drug: Bedaquiline, Delamanid, Moxifloxacin
- Arm5(D800-BD) (Experimental): Participants receive the following medication for the duration of 16weeks together with food.
  * Delpazolid : Will be dosed 800 mg orally twice daily
  * Bedaquiline: will be dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid: will be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin: will be dosed as per the licensed dose: 400 mg orally once daily
  Interventions: Drug: Delpazolid; Drug: Bedaquiline, Delamanid, Moxifloxacin

INTERVENTIONS:
Drug: Delpazolid — Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Other Names: LCB01-0371
  Arms: Arm2(D400); Arm3(D800-OD); Arm4(D1200); Arm5(D800-BD)
Drug: Bedaquiline, Delamanid, Moxifloxacin — These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
  Other Names: BDM

SUMMARY:
This trial is to describe the safety, tolerability and exposure-toxicity relationship of Depazolid given over 16 weeks, in combination with standard-dose Bedaquiline, Delamanid and Moxifloxacin, compared to standard-dose Bedaquiline, Delamanid and Moxifloxacin alone

DETAILED DESCRIPTION:
This will be an open label Phase IIb dose-finding, randomized, controlled study with a duration of 16 weeks of experimental therapy of Delpazolid(DZD) - Bedaquiline/Delamanid/ Moxifloxacin (BDM) in adult patients with newly diagnosed, smear positive, uncomplicated, drug sensitive pulmonary tuberculosis (TB) to evaluate the safety, efficacy, tolerability, pharmacokinetics and exposure/response-relationship of different doses of delpazolid in combination with bedaquiline, delamanid and moxifloxacin.

Participants will be randomized to one of five arms containing BDM standard dose with different doses of DZD.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures including HIV testing.
2. Male or female, aged between 18 and 65 years, inclusive.
3. Body weight between 40 and 90 kg, inclusive.
4. Newly diagnosed, previously untreated, drug susceptible pulmonary TB: presence of MTB complex and rapid molecular tests result confirming susceptibility to RIF and INH such as GeneXpert and/or HAIN MTBDR plus.
5. A chest X-ray (no older than 2 weeks) which, in the opinion of the Investigator, is consistent with TB.
6. Sputum positive on microscopy from concentrated sputum for acid-fast bacilli on at least one sputum sample (at least 1+ on the IUATLD/WHO scale).
7. The participant is willing to forgo consumption of foods high in tyramine for the period of taking study medication (See Appendix, section 20.2, page 92).
8. The participant is either unable to conceive/father children AND/OR his/her partner is unable to conceive/father children AND/OR they will consent to be using effective methods of contraception when engaging in heterosexual intercourse, as defined below:

   a. Non-childbearing potential: i. Female participant/sexual partner of male participant: Bilateral oophorectomy, and/or hysterectomy or bilateral tubal ligation more than 12 months ago and/or has been postmenopausal with a history of no menses for at least 12 consecutive months ii. Male participant/sexual partner of female participant: Vasectomised or has had a bilateral orchidectomy minimally three months prior to screening iii. Male participants having a pregnant female partner or a male sexual partner: At least one barrier method has to be used in this case. b. Effective contraception methods: i. Female participants: Two methods, including methods that the patient's sexual partner(s) use. At least one must be a barrier method. Contraception must be practised for at least until 12 weeks after the last dose of DZD. ii. Male participants: Two methods, including methods that the patient's female sexual partner(s) use. At least one must be a barrier method. Effective contraception must be ensured for at least 16 weeks after the last dose of DZD.

Note: hormone-based contraception alone may not be reliable when taking RIF during continuation phase; therefore, hormone-based contraceptives alone cannot be used by female participants/female partners of male participants to prevent pregnancy.

Exclusion Criteria:

1. Circumstances that raise doubt about free, unconstrained consent to study participation (e.g. prisoner or mentally handicapped person)
2. Poor general condition where delay in treatment cannot be tolerated or death within four months is likely.
3. Poor social condition which would make it unlikely that the patient would be able to complete follow-up
4. The patient is pregnant or breast-feeding.
5. The patient is infected with HIV with a CD4 count <220 cells/mm3. If >220 cells/mm3, patients will be included only if any of the following is applicable:

   * The patient is antiretroviral (ARV) naïve and able to postpone commencing HIV treatment for 2 months after the trial has started and then restrict regimens to those containing dolutegravir (see section 12.6.2 on ARVs) or The patient is ARV experienced (has been on ARV´s a minimum of 5 months) and able to switch to a dolutegravir-based regimen.
   * The patient is treated with nucleosidic reverse transcriptase inhibitors (are permitted as concomitant medication).
   * The patient is treated with protease inhibitors as part of antiretroviral treatment regimens, which will be stopped at least 3 days before the start of study treatment (WK01, day1) for a patient to be eligible.
   * The patient is treated with Efavirenz as part of antiretroviral treatment regimens which would have to be stopped 14 days before the start of study treatment (WK00, Day 01) for a patient to be eligible.
6. The patient has a known intolerance to any of the study drugs or concomitant disorders or conditions for which study drugs or standard TB treatment are contraindicated
7. The patient has a history of, or current evidence of clinically relevant cardiovascular metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or any other condition that will influence treatment response, study adherence or survival in the judgement of the investigator, especially:

   1. Neuropathy, or significant psychiatric disorder like depression or schizophrenia; especially if treatment for those has ever been required or is anticipated to be required
   2. Clinically significant evidence of extra-pulmonary TB (e.g. miliary TB, TB meningitis, but not limited lymph node involvement)
   3. Serious lung conditions other than TB, or significant respiratory impairment in the discretion of the investigator
   4. Any diabetes mellitus
   5. Cardiovascular disease such as myocardial infarction, heart failure, coronary heart disease, arrhythmia, tachyarrhythmia, or pulmonary hypertension
   6. Arterial hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure of ≥90 mmHg on two occasions during screening).
   7. Long QT syndrome or family history of long QT syndrome or sudden death of unknown or cardiac-related cause
   8. Alcohol or other drug abuse that is sufficient to significantly compromise the safety or cooperation of the patient, that includes substances prohibited by the protocol or has led to significant organ damage at the discretion of the investigator.
8. Any of the following laboratory findings at screening:

   1. Serum amino aspartate transferase (AST) and/or alanine aminotransferase (ALT) >3x the upper limit of normal (ULN),
   2. Serum alkaline phosphatase or y-glutamyl transferase > 2.5x the ULN,
   3. Serum total bilirubin level >1.5x the ULN
   4. Estimated creatinine clearance (eCrCl; using the Cockroft and Gault formula [57] lower than 30 ml/min
   5. Serum albumin < 2.8 mg/dl
   6. Haemoglobin level <7.0 g/dl
   7. Platelet count <50,000/mm3
   8. Serum potassium below the lower level of normal for the laboratory
   9. Blood glucose at screening of less than 70mg/dL (3.9mmol/L)
9. ECG findings in the screening ECG: (one or more):

   1. QTcF of >0.450 s
   2. Atrioventricular (AV) block with PR interval > 0.20 s,
   3. QRS complex > 120 milliseconds
   4. Any other changes in the ECG that are clinically relevant as per discretion of the investigator
10. Restricted medication:

    1. Treatment with any other investigational drug within 1 month prior to enrolment or enrolment into other clinical (intervention) trials during participation.
    2. Previous anti-TB treatment with drugs active against MTB within the last 3 months prior to screening.
    3. Unable or unwilling to abide by the requirements regarding restricted medication or have taken restricted medication as described under section 12.6, page 58. Restricted medication includes the following drug classes:

       * Anti-TB drugs other than study drugs
       * Medication that lowers the threshold for epileptic seizures
       * Medication that prolongs the QTc interval
       * Drugs that affect monoaminooxidase or serotonin metabolism
       * CYP 450 inhibitors or inducers, including grapefruit containing foods / beverages and St. John's Wort

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- South Africa (2):
  - The Aurum Institute Tembisa Clinical Research Centre, Tembisa, Gauteng
  - Clinical HIV Research Unit (CHRU) University of the Witwatersrand, Johannesburg
- Tanzania (3):
  - Ifakara Health Institute, Bagamoyo
  - National Institute for Medical Research (NIMR-MMRC), Mbeya
  - Ki'bongoto Infectious Disease Hospital (KIDH) Kilimanjaro Clinical Research Institute (KCRI), Moshi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual patient data, that underlie the results in published article(s) based on data from the trial which including text, tables, figures will be presented to various stakeholders. This reported will be presented to various stakeholder during various forums or meetings. First esults will be disclosed to participants, staff and our site Community Advisory Board. Thereafter we would invite several stakeholders from the community or visit their establishments to review study results. Simultaneously, the studying findings report will be sent to the various regulatory authorities, including the National Department of Health (NDoH). With NDoH and its divisions we will establish needs for further engagement and suggestions for policy or programmatic changes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: PD will be provided 1 - 2 years after and up to 5 years after the publication of the article on the results of the trial
Access Criteria: IPD access will be provided for analyses of related to the aims of research described in the protocol and for individual patient data meta-analyses to researchers who provide a methodologically sound proposal to yhlee@ligachembio.com

REFERENCES:
- [Result] Minja LT, van der Feltz I, Manyama C, Mpagama S, Mhimbira F, Norena I, Sebe M, Rassool M, Wallis RS, Ntinginya N, Liyoyo A, Mbeya B, Wagnerberger L, Zumba T, Peter DD, Makkan H, Sloan DJ, Brake LT, Schildkraut JA, Aarnoutse R, McHugh TD, Wildner L, Boeree MJ, Geiter L, Cho YL, Aldana BH, Phillips PPJ, Hoelscher M, Svensson EM, Heinrich N; PanACEA consortium. Delpazolid in combination with bedaquiline, delamanid, and moxifloxacin for pulmonary tuberculosis (PanACEA-DECODE-01): a prospective, randomised, open-label, phase 2b, dose-finding trial. Lancet Infect Dis. 2025 Nov;25(11):1219-1229. doi: 10.1016/S1473-3099(25)00289-0. Epub 2025 Jul 8. PMID 40645198
- [Derived] Dierig A, Hoelscher M, Schultz S, Hoffmann L, Jarchow-MacDonald A, Svensson EM, Te Brake L, Aarnoutse R, Boeree M, McHugh TD, Wildner LM, Gong X, Phillips P, Minja LT, Ntinginya N, Mpagama S, Liyoyo A, Wallis RS, Sebe M, Mhimbira FA, Mbeya B, Rassool M, Geiter L, Cho YL, Heinrich N. A phase IIb, open-label, randomized controlled dose ranging multi-centre trial to evaluate the safety, tolerability, pharmacokinetics and exposure-response relationship of different doses of delpazolid in combination with bedaquiline delamanid moxifloxacin in adult subjects with newly diagnosed, uncomplicated, smear-positive, drug-sensitive pulmonary tuberculosis. Trials. 2023 Jun 6;24(1):382. doi: 10.1186/s13063-023-07354-5. PMID 37280643

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was initiated on 28 October 2021 (first signed informed consent) with the date of last participant who completed last study visit on 04 Sep 2023.
  A total of 156 participants were screened. Of these, 76 participants were randomized to 1 of 5 arms, and subsequently received at least 1 dose of the study drug. The remaining 80 participants were considered to have been screen failures.
Groups:
- Arm1(D0): Participants received the following medication for the duration of 16 weeks together with food.
  * Delpazolid was not administered
  * Bedaquilin was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm2(D400): Participants received the following medication for the duration of 16 weeks together with food.
  * Delpazolid was dosed 400 mg orally once daily
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm3(D800-OD): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was dosed 800 mg orally once daily
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm4(D1200): Participants received the following medication for the duration of 16 weeks together with food.
  * Delpazolid was dosed 1200 mg orally once daily
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm5(D800-BD): Participants received the following medication for the duration of 16 weeks together with food.
  * Delpazolid was dosed 800 mg orally twice daily
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
Period: Overall Study
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Started (Randomized) | 15 | 15 | 15 | 16 | 15
Received ≥ 1 Dose of Study Drug | 15 | 15 | 15 | 16 | 15
Completed | 15 | 15 | 13 | 16 | 14
Not Completed | 0 | 0 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population and Safety Population
Groups:
- Arm1(D0): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was not administered
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was be dosed as per the licensed dose: 400 mg orally once daily
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm2(D400): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was dosed 400 mg orally once daily
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was be dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm4(D1200): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was be dosed 1200 mg orally once daily
  * Bedaquiline was be dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was be dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm5(D800-BD): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was be dosed 800 mg orally twice daily
  * Bedaquiline was be dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was be dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was be dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Total: Total of all reporting groups
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD) | Total
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.3) | 39.7 (9.0) | 35.1 (11.3) | 34.1 (7.1) | 33.3 (8.4) | 35.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 7 | 4 | 16
  Male | 13 | 15 | 12 | 9 | 11 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 15 | 14 | 16 | 15 | 74
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 15 | 15 | 16 | 15 | 76
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 18.2 (1.8) | 18.8 (2.1) | 20.0 (3.8) | 20.2 (3.0) | 20.0 (3.5) | 19.5 (3.0)
HIV status [Count of Participants; unit: Participants]
  Negative | 13 | 14 | 12 | 13 | 13 | 65
  Positive | 2 | 1 | 3 | 3 | 2 | 11
GeneXpert CT results [Count of Participants; unit: Participants]
  < 16 ; high bacili (TB) load | 3 | 3 | 3 | 3 | 3 | 15
  ≥ 16 ; low bacili (TB) load | 12 | 12 | 12 | 13 | 12 | 61

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome : Proportion of Patients Experiencing Adverse Event
Description: Participants with ≥ 1 TEAE, by severity, related Adverse events: possibly, probably, or definitely related to study drugs
Time Frame: week0 - week52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Arm1(D0): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was not administered
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm2(D400): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was dosed 400 mg orally once daily
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm4(D1200): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was dosed 1200 mg orally once daily
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
- Arm5(D800-BD): Participants receive the following medication for the duration of 16 weeks together with food.
  * Delpazolid was dosed 800 mg orally twice daily
  * Bedaquiline was dosed as per the licensed dose: 400 mg orally once daily for the first 14 days, then 200 mg three times a week.
  * Delamanid was dosed as per the licensed dose: 200 mg orally twice daily doses of 100 mg.
  * Moxifloxacin was dosed as per the licensed dose: 400 mg orally once daily
  Delpazolid: Delpazolid is not licensed yet. Current experience in humans upto Phase IIA. Dose according to randomization to dosing arms 2-5.
  Bedaquiline, Delamanid, Moxifloxacin: These three licensed drugs form the backbone of a new regimen to which delpazolid is added in arms 2-5.
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
Participants
  TEAE (total) | 8 | 7 | 7 | 6 | 9
  Grade 1 (mild) | 4 | 3 | 0 | 0 | 1
  Grade 2 (moderate) | 4 | 4 | 5 | 5 | 7
  Grade 3 (severe) | 0 | 0 | 1 | 1 | 3
  Grade 4 (life-threatening) | 0 | 0 | 2 | 0 | 0
  Unrelated | 5 | 3 | 6 | 3 | 6
  Unlikely related | 0 | 1 | 1 | 1 | 1
  Possibly related | 2 | 1 | 0 | 1 | 4
  Probably related | 0 | 1 | 1 | 1 | 0
  Definitely related | 1 | 1 | 0 | 0 | 0
  SAE- Grade 3 (severe) | 0 | 0 | 0 | 0 | 2
  SAE-Grade 4 (life-threatening) | 0 | 0 | 1 | 0 | 0
  DZD-unrelated SAEs | 0 | 0 | 1 | 0 | 0
  DZD-related SAEs | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Efficacy Outcome: Exposure-response Analysis With TTP (Time to Positive)_AUC0-24
Description: The efficacy of DZD was evaluated by measuring the change in mycobacterial load over time on treatment as quantified by TTP (Time to positive) in BD MGIT960® liquid culture described by non linear mixed effects methodology. A population PK model was developed using NONMEM version 7.4.1. DZD PK is well-described by a two-compartment model with first-order absorption, first-order elimination and a proportional residual error. The final model included allometric scaling based on FFM.
Time Frame: Week 0 - Week 16
Population: Intent to Treat Population; all randomized participants in the groups to which they were randomly assigned and who have taken at least one dose of study treatment.
Measure: Median (Full Range); unit: mg/L*h
Groups:
- Arm1(D0): BDM group
  * Bedaquiline
  * Delamanid
  * Moxifloxacin
- Arm2(D400): BDM + delpazolid 400 mg QD group
- Arm3(D800-OD): BDM + delpazolid 800 mg QD group
- Arm4(D1200): BDM + delpazolid 1200 mg QD group
- Arm5(D800-BD): BDM + delpazolid 800 mg BID group
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
mg/L*h | NA [NA to NA] — Delpazolid is not administered in this arm. | 10.1 [6.86 to 20.4] | 28.6 [15.1 to 76.7] | 47.0 [11.8 to 94.0] | 68.5 [28.8 to 198]

3. Primary Outcome: Efficacy Outcome: Exposure-response Analysis With TTP (Time to Positive)_Cmax
Description: as for outcome 2
Time Frame: Week 0 - Week 16
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/L
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
mg/L | NA [NA to NA] — Delpazolid is not administered in this arm. | 3.78 [2.92 to 4.45] | 7.72 [5.78 to 13.9] | 13.7 [9.56 to 19.7] | 9.16 [7.56 to 13.4]

4. Primary Outcome: Efficacy Outcome: Exposure-response Analysis With TTP (Time to Positive)_Cmin
Description: as for outcome 2
Time Frame: Week 0 - Week 16
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/L
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
mg/L | NA [NA to NA] — Delpazolid is not administered in this arm. | 0.00296 [0.000437 to 0.459] | 0.00948 [0.000439 to 0.810] | 0.00240 [0.000215 to 0.291] | 0.00400 [0.000157 to 0.564]

5. Secondary Outcome: Efficacy Outcome: BD MGIT960® Liquid Media Culture Results
Description: Summary of Changes in Mycobacterial Load Over Time on Treatment as Quantified by Time to Positivity in BD MGIT960® Liquid Media - Intent to Treat Population Sputum samples were collected for BD MGIT960® Liquid Media culture at all time points during the treatment and follow-up phases, and this table shows culture results, which are reported as: Positive, Negative, Contaminated, Missing.
  Note: Contaminated cultures are shown as contaminated for the purpose of the overall result but are counted as missing for calculating summary statistics. The data recorded as 'Positive for MTB Complex with Contamination' are included as 'Positive' for MGIT result. However, the data from mean and median calculations for TTP (Time to positive) due to contamination.
Time Frame: Week 0 - Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
Participants
  Week 0: Positive | 15 | 15 | 15 | 16 | 15
  Week 0: Negative | 0 | 0 | 0 | 0 | 0
  Week 0: Contaminated | 0 | 0 | 0 | 0 | 0
  Week 0: Missing | 0 | 0 | 0 | 0 | 0
  Week 1: Positive | 15 | 14 | 15 | 15 | 15
  Week 1: Negative | 0 | 1 | 0 | 1 | 0
  Week 1: Contaminated | 0 | 0 | 0 | 0 | 0
  Week 1: Missing | 0 | 0 | 0 | 0 | 0
  Week 2: Positive | 15 | 14 | 14 | 16 | 15
  Week 2: Negative | 0 | 1 | 1 | 0 | 0
  Week 2: Contaminated | 0 | 0 | 0 | 0 | 0
  Week 2: Missing | 0 | 0 | 0 | 0 | 0
  Week 3: Positive | 15 | 13 | 12 | 15 | 15
  Week 3: Negative | 0 | 2 | 1 | 0 | 0
  Week 3: Contaminated | 0 | 0 | 0 | 1 | 0
  Week 3: Missing | 0 | 0 | 2 | 0 | 0
  Week 4: Positive | 13 | 13 | 13 | 14 | 12
  Week 4: Negative | 2 | 2 | 1 | 2 | 3
  Week 4: Contaminated | 0 | 0 | 0 | 0 | 0
  Week 4: Missing | 0 | 0 | 1 | 0 | 0
  Week 5: Positive | 14 | 12 | 11 | 13 | 12
  Week 5: Negative | 1 | 3 | 2 | 3 | 3
  Week 5: Contaminated | 0 | 0 | 0 | 0 | 0
  Week 5: Missing | 0 | 0 | 2 | 0 | 0
  Week 6: Positive | 9 | 9 | 12 | 10 | 12
  Week 6: Negative | 5 | 6 | 2 | 6 | 3
  Week 6: Contaminated | 1 | 0 | 0 | 0 | 0
  Week 6: Missing | 0 | 0 | 1 | 0 | 0
  Week 7: Positive | 9 | 8 | 5 | 8 | 8
  Week 7: Negative | 6 | 7 | 9 | 8 | 7
  Week 7: Contaminated | 0 | 0 | 0 | 0 | 0
  Week 7: Missing | 0 | 0 | 1 | 0 | 0
  Week 8: Positive | 6 | 6 | 5 | 2 | 7
  Week 8: Negative | 9 | 9 | 9 | 13 | 7
  Week 8: Contaminated | 0 | 0 | 0 | 1 | 1
  Week 8: Missing | 0 | 0 | 1 | 0 | 0
  Week 9: Positive | 5 | 4 | 3 | 3 | 2
  Week 9: Negative | 10 | 11 | 11 | 13 | 11
  Week 9: Contaminated | 0 | 0 | 0 | 0 | 1
  Week 9: Missing | 0 | 0 | 1 | 0 | 1
  Week 10: Positive | 4 | 3 | 1 | 3 | 3
  Week 10: Negative | 10 | 12 | 12 | 13 | 11
  Week 10: Contaminated | 1 | 0 | 1 | 0 | 1
  Week 10: Missing | 0 | 0 | 1 | 0 | 0
  Week 11: Positive | 3 | 2 | 1 | 1 | 2
  Week 11: Negative | 11 | 12 | 13 | 14 | 13
  Week 11: Contaminated | 1 | 1 | 0 | 1 | 0
  Week 11: Missing | 0 | 0 | 1 | 0 | 0
  Week 12: Positive | 2 | 0 | 0 | 0 | 2
  Week 12: Negative | 12 | 15 | 14 | 16 | 13
  Week 12: Contaminated | 1 | 0 | 0 | 0 | 0
  Week 12: Missing | 0 | 0 | 1 | 0 | 0
  Week 13: Positive | 0 | 0 | 0 | 0 | 3
  Week 13: Negative | 15 | 15 | 14 | 15 | 12
  Week 13: Contaminated | 0 | 0 | 0 | 1 | 0
  Week 13: Missing | 0 | 0 | 1 | 0 | 0
  Week 14: Positive | 1 | 0 | 0 | 0 | 2
  Week 14: Negative | 13 | 15 | 12 | 14 | 11
  Week 14: Contaminated | 1 | 0 | 2 | 2 | 2
  Week 14: Missing | 0 | 0 | 1 | 0 | 0
  Week 15: Positive | 1 | 0 | 0 | 0 | 1
  Week 15: Negative | 14 | 15 | 13 | 16 | 14
  Week 15: Contaminated | 0 | 0 | 1 | 0 | 0
  Week 15: Missing | 0 | 0 | 1 | 0 | 0
  Week 16: Positive | 0 | 0 | 0 | 0 | 1
  Week 16: Negative | 14 | 15 | 14 | 16 | 14
  Week 16: Contaminated | 1 | 0 | 0 | 0 | 0
  Week 16: Missing | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Efficacy Outcome: Changes in Mycobacterial Load Over Time on Treatment as Quantified by Time to Positivity in BD MGIT960® Liquid Media
Description: The efficacy of DZD was evaluated by measuring the change in mycobacterial load over time on treatment as quantified by time to positivity (TTP) in BD MGIT 960® liquid culture described by nonlinear mixed-effects methodology. Sputum samples were collected for BD MGIT960® Liquid Media culture at all time points during the treatment and follow-up phases, and this table shows TTP results.
Time Frame: Week 0 - Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
days
  Week 0 | 5.6 (2.2) | 6.5 (4.1) | 7.2 (5.7) | 8.0 (9.0) | 5.9 (2.2)
  Week 1 | 10.9 (3.2) | 13.0 (8.9) | 10.1 (3.8) | 11.1 (8.8) | 9.6 (3.3)
  Week 2 | 13.3 (4.3) | 16.9 (9.9) | 15.4 (8.6) | 13.7 (7.8) | 12.2 (3.7)
  Week 3 | 16.6 (6.5) | 18.0 (11.8) | 16.0 (8.4) | 14.2 (6.4) | 15.7 (8.2)
  Week 4 | 19.1 (10.4) | 18.3 (10.3) | 18.7 (8.1) | 21.2 (10.1) | 19.8 (12.1)
  Week 5 | 23.6 (9.2) | 24.4 (11.0) | 23.3 (10.1) | 25.3 (10.4) | 23.8 (10.8)
  Week 6 | 27.3 (11.9) | 29.7 (11.4) | 2.74 (8.4) | 27.9 (12.1) | 26.9 (10.3)
  Week 7 | 30.8 (11.7) | 31.6 (10.9) | 35.1 (9.7) | 33.6 (10.9) | 30.9 (12.5)
  Week 8 | 33.3 (12.0) | 36.6 (8.9) | 36.3 (9.7) | 39.4 (7.5) | 33.2 (11.1)
  Week 9 | 35.8 (10.3) | 37.7 (9.7) | 38.0 (8.3) | 37.0 (10.9) | 38.8 (7.8)
  Week 10 | 36.4 (10.1) | 37.8 (9.1) | 40.5 (5.4) | 39.3 (7.3) | 39.7 (5.5)
  Week 11 | 36.6 (11.5) | 40.1 (5.2) | 40.9 (4.3) | 41.4 (2.4) | 38.5 (9.4)
  Week 12 | 38.5 (9.3) | 42.0 (0) | 42.0 (0) | 42.0 (0) | 40.0 (6.1)
  Week 13 | 42.0 (0) | 42.0 (0) | 42.0 (0) | 42.0 (0) | 39.2 (7.3)
  Week 14 | 39.9 (8.0) | 42.0 (0) | 42.0 (0) | 42.0 (0) | 39.4 (7.8)
  Week 15 | 39.7 (8.9) | 42.0 (0) | 42.0 (0) | 42.0 (0) | 40.0 (7.8)
  Week 16 | 42.0 (0) | 42.0 (0) | 42.0 (0) | 42.0 (0) | 40.0 (7.7)

7. Secondary Outcome: Efficacy Outcome: Loewenstein-Jensen Solid Media Culture Results
Description: Summary of Changes in Mycobacterial Load Over Time on Treatment as Quantified by Time to Culture Conversion in Loewenstein-Jensen Solid Media - Intent-to-Treat Population Sputum samples were collected for Loewenstein-Jensen Solid Media culture at at Week 0, Week 8, Week 12, Week 6 during the treatment and follow-up phases, and this table shows culture results, which are reported as: Positive, Negative, Contaminated, Missing.
Time Frame: Week 0 - Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
Participants
  Week 0: Positive | 14 | 15 | 15 | 16 | 15
  Week 0: Negative | 1 | 0 | 0 | 0 | 0
  Week 0: Contaminated | 0 | 0 | 0 | 0 | 0
  Week 0: Missing | 0 | 0 | 0 | 0 | 0
  Week 8: Positive | 4 | 2 | 3 | 1 | 3
  Week 8: Negative | 11 | 12 | 11 | 15 | 12
  Week 8: Contaminated | 0 | 1 | 0 | 0 | 0
  Week 8: Missing | 0 | 0 | 1 | 0 | 0
  Week 12: Positive | 2 | 0 | 0 | 0 | 1
  Week 12: Negative | 13 | 15 | 14 | 16 | 14
  Week 12: Contaminated | 0 | 0 | 0 | 0 | 0
  Week 12: Missing | 0 | 0 | 1 | 0 | 0
  Week 16: Positive | 0 | 0 | 0 | 0 | 1
  Week 16: Negative | 14 | 15 | 14 | 16 | 14
  Week 16: Contaminated | 1 | 0 | 0 | 0 | 0
  Week 16: Missing | 0 | 0 | 1 | 0 | 0

8. Secondary Outcome: Efficacy Outcome: The Proportion Converted by Day Corresponding to End of Each Week
Description: Culture conversion was defined as 2 negative cultures without an intervening positive culture. Time was measured as time on treatment until the first negative culture (up to Week 16 Visit).
  'Converted by Week x' shows proportion converted by day corresponding to end of each week, e.g., Week 2 = Day 14.
Time Frame: Week 0 - Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
percentage of participants
  Week 0 | 0 | 0 | 0 | 0 | 0
  Week 2 | 0 | 6.7 | 6.7 | 0 | 0
  Week 3 | 0 | 6.7 | 6.7 | 0 | 0
  Week 4 | 6.7 | 6.7 | 13.8 | 6.2 | 13.3
  Week 5 | 6.7 | 20.0 | 13.8 | 18.8 | 13.3
  Week 6 | 33.3 | 40.0 | 21.0 | 37.5 | 13.3
  Week 7 | 40.0 | 46.7 | 64.1 | 43.8 | 40.0
  Week 8 | 60.0 | 73.3 | 64.1 | 75.0 | 46.7
  Week 9 | 60.0 | 86.7 | 78.5 | 87.5 | 73.3
  Week 10 | 66.7 | 86.7 | 92.8 | 87.5 | 80.0
  Week 11 | 73.3 | 86.7 | 92.8 | 93.8 | 86.7
  Week 12 | 80.0 | 100 | 100 | 100 | 86.7
  Week 13 | 93.3 | 100 | 100 | 100 | 86.7
  Week 14 | 93.3 | 100 | 100 | 100 | 86.7
  Week 15 | 93.3 | 100 | 100 | 100 | 93.3
  Week 16 | 93.3 | 100 | 100 | 100 | 93.3

9. Secondary Outcome: Efficacy Outcome: Time to Culture Conversion
Description: Time to culture conversion was defined as 2 negative cultures without an intervening positive culture. Time was measured as time on treatment until the first negative culture (up to Week 16 Visit).
Time Frame: Week 0 - Week 16
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
Days | 56.0 [42.0 to 84.0] | 56.0 [42.0 to 63.0] | 59.0 [49.0 to 63.0] | 56.0 [42.0 to 59.5] | 63.0 [49.0 to 70.0]

10. Secondary Outcome: Efficacy Outcome : Relapse or Reinfection
Description: A participant was positive for relapse or reinfection if they converted to culture negative by Week 8 and had 2 consecutive positive cultures after Week 16 of randomization, without an intervening negative.
Time Frame: Week0 - Week52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Arm1(D0): BDM alone
  * Bedaquiline
  * Delamanid
  * Moxifloxacin
- Arm2(D400): BDM + delpazolid 400 mg QD
  * Delpazolid 400 mg QD
  * Bedaquiline
  * Delamanid
  * Moxifloxacin
- Arm3(D800-OD): BDM + delpazolid 800 mg QD
  * Delpazolid 800 mg QD
  * Bedaquiline
  * Delamanid
  * Moxifloxacin
- Arm4(D1200): BDM + delpazolid 1200 mg QD
  * Delpazolid 1200 mg QD
  * Bedaquiline
  * Delamanid
  * Moxifloxacin
- Arm5(D800-BD): BDM + delpazolid 800 mg BIDD
  * Delpazolid 800 mg BID
  * Bedaquiline
  * Delamanid
  * Moxifloxacin
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 15
Participants
  Conversion by Week 8 and no positive culture past week 12 | 9 | 11 | 10 | 12 | 5
  Conversion by Week 8 and positive culture past week 12 | 0 | 0 | 0 | 0 | 2
  Did not convert by Week 8 | 6 | 4 | 5 | 4 | 8
  Relapsed or reinfected | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Week 0 to Week 52
Arm/Group | Arm1(D0) | Arm2(D400) | Arm3(D800-OD) | Arm4(D1200) | Arm5(D800-BD)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/15 | 0/16 | 2/15
Other Adverse Events (participants affected / at risk) | 8/15 | 7/15 | 7/15 | 6/16 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm1(D0) (N=15) | Arm2(D400) (N=15) | Arm3(D800-OD) (N=15) | Arm4(D1200) (N=16) | Arm5(D800-BD) (N=15)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm1(D0) (N=15) | Arm2(D400) (N=15) | Arm3(D800-OD) (N=15) | Arm4(D1200) (N=16) | Arm5(D800-BD) (N=15)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Gamma glutamyl transferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04550832/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT04550832/SAP_001.pdf